CLINICAL TRIAL: NCT06737991
Title: Effects of Chest Expansion Exercises on Thoracic Expansion and VO2 Max in Children With Chest Burn
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REC/RCR/AHS/24/Kashaf
Record Dates: First submitted 2024-11-12; First posted 2024-12-17 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Burns Multiple
MeSH Terms: interventions — Range of Motion, Articular

STUDY DESIGN:
Intervention Model Description: On the group of children with chest burn, thoracic expansion exercises will be applied and VO2 Max will be monitored.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Quasi Group (Experimental): A group of 33 children of age 5-10 years with chest burn. The techniques include deep breathing with shoulder abduction, deep breathing and relaxing with hip external rotation with slight knee flexion, floor polishing motion; rounded hands to draw small circles on the floor etc.
  Interventions: Other: Range of motion exercises

INTERVENTIONS:
Other: Range of motion exercises — Range of motion Exercises, soft tissue massage, positioning to prevent pressure sores, stretch pole for 20 minutes

SUMMARY:
Burns are injuries to the skin or tissues caused by heat, electricity, chemicals, friction, or radiation. They can result from flames, hot solids, or liquids. In intensive care, physiotherapy often includes sitting exercises, passive motions, and active training, which are essential for recovery after burns. This study aims to evaluate the impact of chest expansion exercises using a stretch pole on chest expansion and VO2 max in children with chest burns. Conducted as a quasi-experimental study at Jinnah Burn Centre in Lahore, it will involve 33 participants selected through non-probability convenience sampling. Data collection will span six months. Thoracic expansion will be measured with an inch tape, and VO2 max will be calculated using a specific formula. Routine physiotherapy, including range of motion exercises and soft tissue massage, will be administered alongside chest expansion exercises for 20 minutes daily, five days a week, over three weeks.

DETAILED DESCRIPTION:
Burns are a kind of injury that can occur to the skin or other tissues. Acute trauma can be brought on by heat, electricity, chemicals, friction, radiation, or other factors. Burns are a kind of injury that can occur to the skin or other tissues. Acute trauma can be brought on by heat, electricity, chemicals, friction, radiation, or other factors. Burn are many types of burn Flames (flame burns), hot solids (contact burns), or hot liquids (scalds). Sitting out of bed, passive motions, and active/assisted exercises were frequent physiotherapy therapies in the intensive care unit. After a burn injury, exercise training serves as a significant and useful technique for achieving physical health. The objective of this study is to check the effect of chest expansion exercises by using stretch pole on chest expansion and VO2 max in children with chest burn. This study will be a Quasi-Experimental study .Data will be collected from Jinnah Burn Centre, Lahore. Data will be collected within 6 month from approval date of synopsis. Sample size is 33. Non-probability convenience sampling technique will be used in this study. Thoracic expansion will be measured by inch tape and vo2 max will be calculated by using a formula. Routine physiotherapy will be provided to the subjects routinely with chest expansion exercises. In routine physiotherapy, Range of motion exercises, Soft tissue massage, positioning to prevent the pressure sores will be provided for almost 20 minutes. The chest expansion exercises will be provided to the patients by using stretch pole for 20 minutes. All the interventions will be given to patients for 5 days in a week on daily basis for 3 weeks

ELIGIBILITY:
Inclusion Criteria:

* Age: 5- 10 years.
* Children with mild to moderate chest burn.
* Children with decreased mobility due to chest burn.

Exclusion Criteria:

* Chest burns with any post-burn complications,
* Neurological impairments,
* Contracture due to immobility,
* Infection due to chest burn.

Ages: 5 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 33 (Estimated)
Dates: Start 2024-06-12 (Actual); Primary Completion 2024-10-10 (Actual); Study Completion 2024-12-17 (Estimated)

PRIMARY OUTCOMES:
Chest Expansion | 6 months
  Chest expansion refers to the increase in chest cavity size during breathing, essential for effective lung function and oxygen intake.
VO2 Max | 6 months
  VO2 max is the maximum amount of oxygen the body can utilize during intense exercise, reflecting aerobic fitness and cardiovascular health.

CONTACTS AND LOCATIONS:
Overall Officials: Kashaf Ahmad, MS*, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kaur D, Sharma N, Samuel AJ. Web-based E-survey in identifying current physiotherapy practices in paediatric burns. Burns. 2023 Sep;49(6):1474-1481. doi: 10.1016/j.burns.2023.01.009. Epub 2023 Jan 25. PMID 36792471